CLINICAL TRIAL: NCT06928454
Title: INFORMED: Brain Health Project for Korean American Dementia Caregivers
Brief Title: Brain Health Project for Korean American Dementia Caregivers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-40879
Record Dates: First submitted 2025-03-31; First posted 2025-04-15 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Caregiving Stress
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Brain Health Project (Experimental): Text messages
  Interventions: Behavioral: Text messages over 8 weeks

INTERVENTIONS:
Behavioral: Text messages over 8 weeks — Learn about ADRD/Prepare as a care partner/Care for yourself/Get support

SUMMARY:
The caregivers of persons with dementia face significant emotional, physical, and financial challenges, particularly among under-resourced communities like Korean Americans, who encounter unique obstacles, including language barriers and limited culturally tailored resources. In this pilot study, the investigators propose the Brain Health Project, which focuses on increasing knowledge of Alzheimer's disease and related dementia and enhancing caregiving skills among Korean American dementia caregivers.

ELIGIBILITY:
Inclusion Criteria:

* age 18 and older
* self-identified as Korean American
* able to read and/or speak English or Korean
* care for a person with undiagnosed or diagnosed dementia for the last 6 months
* have access to a mobile phone to receive text messages

Exclusion Criteria:

* planning a trip out of the United States during the next four months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10-14 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Dementia Knowledge Assessment Tool 2 (DKAT2) | Baseline and through study completion, an average of 9 weeks
  Questions to assess dementia knowledge. The higher the final score, the higher the knowledge about dementia (possible scores: 0 - 21).

CONTACTS AND LOCATIONS:
Overall Officials: Ji Won Choi, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No